CLINICAL TRIAL: NCT06873724
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single Dose Study of the Safety, Tolerability, and Pharmacokinetics of SPY003-207 in Healthy Participants
Brief Title: SPY003-207 in Healthy Volunteers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Spyre Therapeutics, Inc. (Industry)
Collaborators: Altasciences Company Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: SPY003-207-101
Record Dates: First submitted 2025-03-07; First posted 2025-03-13 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SAD Cohorts 1-6 Experimental Arm (Experimental): Participants will receive a single dose of SPY003-207 in a dose escalation format
  Interventions: Drug: SPY003-207
- SAD Cohorts 1-6 Placebo Arm (Placebo Comparator): Participants will receive a single dose of placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: SPY003-207 — Experimental
  Arms: SAD Cohorts 1-6 Experimental Arm
Other: Placebo — Placebo
  Arms: SAD Cohorts 1-6 Placebo Arm

SUMMARY:
This is a Phase 1, randomized, double-blind, placebo-controlled, single dose, first in human safety, tolerability, and pharmacokinetic study of SPY003-207 in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* Willing and able to attend the necessary visits to the CRU, comply with all testing requirements, remain at the study site unit for the duration of the confinement period and return for the outpatient visits

Exclusion Criteria:

* Participation in more than one cohort
* Evidence of clinically significant abnormality or disease
* Known history of illicit drug use or drug abuse, harmful alcohol use or alcoholism, and/or smoking or nicotine-containing product use within 3 months prior to the first dose of study drug
* History of severe allergic reactions or hypersensitivity
* Donation or loss of >1 unit of whole blood within 1 month prior to dosing

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Treatment emergent adverse events | Up to 63 weeks
  Incidence, severity, and causal relationship of TEAEs

SECONDARY OUTCOMES:
Cmax | Up to 63 weeks
  Maximum concentration after a single dose
Tmax | Up to 63 weeks
  Time to reach maximum concentration after a single dose
t1/2 | Up to 63 weeks
  Half life after a single dose
AUC | Up to 63 weeks
  Area under the curve after a single dose
ADA | Up to 63 weeks
  Incidence of anti-drug antibody after a single dose

CONTACTS AND LOCATIONS:
Overall Officials: Deanna Nguyen, MD, Study Chair — Spyre Therapeutics
Locations (1):
- Spyre Site 1, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No